CLINICAL TRIAL: NCT05233462
Title: Height Adjusted Versus Standardized Dose of Bupivacaine in Spinal Anesthesia for Caesarean Delivery - A Randomized Double-blind Interventional Study
Brief Title: Height Adjusted Versus Standardized Dose of Bupivacaine for Spinal Anesthesia
Acronym: RAMCES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 21-0217
Record Dates: First submitted 2022-01-31; First posted 2022-02-10 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Regional Anesthesia Morbidity; Cesarean Section Complications; Local Anesthetic Complication
Keywords: cesarean section; intrathecal anesthesia; bupivacaine; morbidity
MeSH Terms: interventions — EPOCH protocol

STUDY DESIGN:
Intervention Model Description: randomized controlled double blind trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Neither the patient nor the care provider nor the outcome assessor will know the allocation group.
  Bupivacaine syringe will be prepare, according to the protocol, by a separate anesthetist not involved in the care of the patient. The solution in both groups will have the same volume.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Active Comparator): intrathecal administration of a solution containing
  * bupivacaine 10 mg
  * morphine 100 micrograms
  * sufentanil 3 micrograms
  Interventions: Other: standardized dose
- individualized group (Experimental): intrathecal administration of a solution containing
  * bupivacaine 0.05 mg per cm of patient's height
  * morphine 100 micrograms
  * sufentanil 3 micrograms
  Interventions: Other: adjusted dose

INTERVENTIONS:
Other: standardized dose — intrathecal anesthesia with 10 mg of bupivacaine
  Other Names: standardized dose of bupivacaine
  Arms: control group
Other: adjusted dose — intrathecal anesthesia with 0.05 mg of bupivacaine par cm of patient's height
  Other Names: adjusted dose of bupivacaine
  Arms: individualized group

SUMMARY:
General anesthesia during pregnancy is associated with several major risks including unanticipated difficult airway, pulmonary aspiration, and specific anesthetic effects on the newborn. Thus, intrathecal anesthesia is the technique of choice for cesarean section.

Nevertheless, the main side effect of intrathecal anesthesia is arterial hypotension which depend mainly on the dose of local anesthetic administered intrathecally.

To date there is no guidelines nor evidences whic help the anesthetist to precisely estimate the required dose. Most often a "standardized dose" of 8 to 10 mg of bupivacaine is administered. However, some data suggest that a lower dose may be administered resulting in less frequent arterial hypotension. Nevertheless, a well designed randomized study is lacking.

DETAILED DESCRIPTION:
The present controlled randomized double blind trial was designed to compare 2 intrathecal dose of bupivacaine for cesarean section

* a "standard" dose of 10 mg of intrathecal bupivacaine associated with morphine 100 micrograms and sufentanil 3 micrograms
* a height-calculated dose of bupivacaine (0.05 mg per cm of height) on associated with morphine 100 micrograms and sufentanil 3 micrograms

The main outcome is the rate of hypotension defined as a 20% or more decrease in systolic arterial pressure.

Secondary outcomes focused on intrathecal anesthesia efficacy, success or failure and on interventions required to manage arterial hypotension

ELIGIBILITY:
Inclusion Criteria:

* scheduled cesarean section with intrathecal anesthesia
* term pregnancy > 35 weeks
* signed informed consent

Exclusion Criteria:

* unscheduled or emergent cesarean section
* any contra indication to intrathecal anesthesia
* any antihypertensive drug prescribed to control arterial pressure during pregnancy
* pre-eclampsia and eclampsia
* history of Marfan or Ehlers Danlos disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnancy and scheduled cesarean section
Enrollment: 250 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
rate of arterial hypotension | 4 hours since the start of intrathecal bupivacaine administration
  rate of arterial hypotension defined as a 20% or more decrease in systolic arterial pressure as compared with baseline systolic arterial pressure measured at 32 weeks

SECONDARY OUTCOMES:
vasopressor total dose | 4 hours since the start of intrathecal bupivacaine administration
  total dose of vasopressor administered during intrathecal anesthesia
metameric level of intrathecal anesthesia | 4 hours since the start of intrathecal bupivacaine administration
  clinical evaluation of the metameric level obtained during intrathecal anesthesia
lower limb motor block at the end of the caesarean section | 5 min after the end of caesarean section at newborn umbilical cord clamp
  lower limb motor block at the end of the caesarean section using Bromage score
rate of need for general anesthesia | 5 min after the end of caesarean section at newborn umbilical cord clamp
  rate of need for general anesthesia because of intrathecal anesthesia failure or overdose
patient's comfort self evaluation | 4 hours since the start of intrathecal bupivacaine administration
  patient's comfort self evaluation using a verbal rating scale from 0 (uncomfortable) to 10 (totally comfortable)

CONTACTS AND LOCATIONS:
Overall Officials: jean-luc hanouz, Study Chair — University Hospital of Caen
Locations (1):
- Caen University Hospital, Caen, France